CLINICAL TRIAL: NCT06648824
Title: A Phase 1, Open-label, One-Sequence Crossover Study to Assess the Effect of Mitapivat on the Pharmacokinetics of the CYP3A Substrate (Midazolam) in Healthy Participants
Brief Title: Study of How Mitapivat Affects Midazolam Blood Levels in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-027
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
Keywords: AG-348; Mitapivat
MeSH Terms: interventions — mitapivat; Midazolam

STUDY DESIGN:
Intervention Model Description: Single sequence crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mitapivat and Midazolam (Experimental): Participants will receive single oral dose of 2 milligram (mg) midazolam on Day 1 followed by 100 mg mitapivat, orally, twice daily (BID) from Day 3 to 13. On Day 14, participants will receive single oral dose of 2 mg midazolam and 100 mg mitapivat orally, BID. Midazolam will be co-administered with morning mitapivat dose.
  Interventions: Drug: Mitapivat; Drug: Midazolam

INTERVENTIONS:
Drug: Mitapivat — Oral tablets
  Other Names: AG-348; PYRUKYND®; AG-348 sulfate hydrate; Mitapivat sulfate
Drug: Midazolam — Oral syrup

SUMMARY:
The primary purpose of this study is to assess the effect of mitapivat on the single oral dose pharmacokinetics (PK) of midazolam in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Females must not be pregnant or lactating.
* Females of childbearing potential must agree to use contraception.
* Body mass index between 18.0 and 32.0 kilogram per meter square (kg/m^2), inclusive.
* In good health, as determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG) and vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in, and from the physical examination at check-in, as assessed by the investigator or designee.
* Able to comprehend and willing to sign the informed consent form (ICF) and abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, ophthalmological (acute angle closure glaucoma), or psychiatric disorder, as determined by the investigator or designee.
* History of significant hypersensitivity, intolerance, or allergy to any relevant drug compound, food, or other substance (ie, allergy to study intervention or excipients [microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, magnesium stearate, and the Opadry Blue II film-coat [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and FD&C Blue #2]]).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (e.g., cholecystectomy). Uncomplicated appendectomy and hernia repair are allowed.
* Significant acute, new-onset illness (e.g., flu, gastroenteritis) within 2 weeks prior to dosing.
* Confirmed systolic blood pressure >150 or <90 millimeters of mercury (mmHg), diastolic blood pressure >100 or <50 mmHg, or pulse rate >100 or <40 beats per minute (bpm). If any parameter falls outside of the specified range at screening or check-in, 2 repeat measurements will be performed and the participant will be excluded only if the mean of the parameter based on the 3 replicates falls outside of the specified range.
* Clinically significant cardiac history or presence of ECG findings, including any of the following:

  1. Heart rate <40 bpm or >100 bpm
  2. Risk factors for torsades de pointes (e.g., heart failure, cardiomyopathy, or family history of long QT syndrome)
  3. Sick sinus syndrome, second- or third-degree atrioventricular block myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities
  4. QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 millisecond (msec) (healthy male participants) or >470 msec (healthy female participants); if QTcF is >450 msec (males) or >470 msec (females), 2 repeat measurements will be performed and the participant will be excluded only if the mean QTcF based on the 3 replicate ECGs is >450 msec (males) or >470 msec (females).
  5. QRS duration >110 msec, confirmed by manual overread; if value is >110 msec, 2 repeat measurements will be performed and the participant will be excluded only if the mean QRS duration based on the 3 replicate ECGs is >110 msec.
  6. PR interval <120 or >220 msec, confirmed by manual overread; if value is <120 or >220 msec, 2 repeat measurements will be performed and the participant will be excluded only if the mean PR interval based on the 3 replicate ECGs is <120 or >220 msec.
  7. Repeated syncope or vasovagal episodes.
  8. Hypertension, angina, bradycardia (if assessed as clinically significant by the investigator) or severe peripheral arterial circulatory disorders
  9. History of autonomic dysfunction.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Administration of any vaccine within 30 days prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
* Use or intend to use any prescription medications/products, other than non-hormonal contraceptives, within 14 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
* Use or intend to use any slow-release medications/products considered to still be active within 14 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
* Use or intend to use any nonprescription medications/products including vitamins, minerals, high-dose biotin supplements and other supplements, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
* Participation in a clinical study involving administration of an investigational medicinal product (new chemical entity) in the past 30 days or 5 half-lives of that drug (if known) prior to dosing, whichever is longer.
* Has previously completed or withdrawn from this study or any other study investigating mitapivat and has previously received mitapivat.
* Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12-ounce (oz) (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Positive urine drug screen at screening; positive alcohol test result or positive urine drug screen at check-in.
* History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in. Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in and not willing to refrain from consumption of these foods or beverages throughout the study until end of study.
* Consumption of caffeine- or xanthine-containing products within 48 hours prior to check-in and not willing to refrain from consumption of these products while at the study site.
* Consumption of vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussel sprouts, and mustard greens), or charbroiled meat within 7 days prior to dosing and not willing to refrain from consumption of these foods until end of study.
* Receipt of blood products within 2 months prior to check-in.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve Extrapolated From Time Zero to Infinity (AUC0-infinity) of Midazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-t) of Midazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Maximum Observed Plasma Concentration (Cmax) of Midazolam | Pre-dose and at multiple timepoints post-dose up to Day 14

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 Hours Post-dose (AUC0-12) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Maximum Observed Plasma Concentration (Cmax) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Area Under the Plasma Concentration-Time Curve Over a Dosing Interval (Tau) at Steady State (AUC0-tau,ss) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Time to Last Measurable Concentration (tlast) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Time to Reach Maximum Concentration (tmax) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 14
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-infinity) of 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-t) of 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Maximum Observed Plasma Concentration (Cmax) of 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Metabolite-to-Parent Ratio of Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-infinity) for Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Metabolite-to-Parent Ratios of Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-t) for Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Metabolite-to-Parent Ratio of Maximum Observed Plasma Concentration (Cmax) for Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Percentage of Area Under the Concentration-Time Curve Due to Extrapolation From the Last Quantifiable Concentration to Infinity (AUC%extrap) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Time to Last Measurable Concentration (tlast) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Time to Reach Maximum Concentration (tmax) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Terminal Elimination Half-Life (t1/2) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Apparent Total Body Clearance (CL/F) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Midazolam and 1'-hydroxymidazolam | Pre-dose and at multiple timepoints post-dose up to Day 14
Number of Participants With Adverse Events (AEs), AEs by Severity, and Relatedness to Study Treatment | Up to Day 24
Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Assessments | Baseline up to Day 24
Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Parameters | Baseline up to Day 14
Number of Participants With Clinically Significant Change From Baseline in Vital Signs Parameters | Baseline up to Day 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Fortrea Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No